CLINICAL TRIAL: NCT05593432
Title: A Randomized, Double-Blind, Vehicle-Controlled Study of the Efficacy and Safety of Ruxolitinib Cream in Participants With Cutaneous Lichen Planus
Brief Title: A Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Participants With Cutaneous Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-216
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-08

CONDITIONS: Cutaneous Lichen Planus
Keywords: Lichen Planus; Skin Diseases; 18424; Ruxolitinib; topical cream
MeSH Terms: conditions — Lichen Planus; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Study will include a 16 week double-blind period followed by a 16 week open-label period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib cream (Experimental): Ruxolitinib 1.5% cream BID for 16 weeks, followed by ruxolitinib cream BID 16-week open-label extension.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle cream
- Vehicle Cream (Placebo Comparator): Vehicle cream BID for 16 weeks, followed by ruxolitinib 1.5% cream BID in a 16-week open-label extension.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB018424 cream
  Arms: Ruxolitinib cream
Drug: Vehicle cream — Vehicle cream is matching in appearance to ruxolitinib cream and is to be applied in the same manner as ruxolitinib cream.

SUMMARY:
The purpose of this study will be to evaluate efficacy and safety of Ruxolitinib cream in participants With Cutaneous Lichen Planus. This is randomized, double-blind, vehicle-controlled (DBVC) study with a DBVC period of 16 weeks followed by an open label period (OLE) period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of LP with predominant cutaneous involvement.
* IGA score of 3 or 4 at screening and baseline.
* Baseline LP-related Itch NRS score ≥ 4.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Concurrent conditions and history of other diseases:

  1. Variants of LP deemed by the investigators to be inappropriate for topical treatment, including but not limited to predominant mucosal (such as oral or vaginal) LP.
  2. Active ongoing inflammatory diseases of the skin other than LP that might confound the evaluation of LP lesions or compromise participant safety.
  3. Any other concomitant skin disorder (eg, generalized erythroderma such as Netherton's syndrome), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of LP lesions or compromise participant safety.
  4. Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, or Wiskott-Aldrich syndrome).
  5. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before baseline.
  6. Active acute bacterial, fungal, or viral skin infection (eg, herpes simplex, herpes zoster, chickenpox, clinically infected AD, or impetigo) within 1 week before baseline.
* Laboratory values outside of the protocol-defined criteria.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.
* Other exclusive criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, Study Director — Incyte Corporation
Locations (24):
- United States (22):
  - Cahaba Dermatology, Birmingham, Alabama
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Wallace of Beverly Hills, Los Angeles, California
  - Northshore Medical Group Dermatology Skokie, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group Llc, Indianapolis, Indiana
  - Delricht Clinical Research-Clinedge-Ppds Baton Rouge, Baton Rouge, Louisiana
  - Delricht Research - Touro Medical Center, New Orleans, Louisiana
  - Dermassociates, Rockville, Maryland
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Jdr Dermatology Research, Las Vegas, Nevada
  - OPTISKIN, New York, New York
  - Bexley Dermatology, Bexley, Ohio
  - Clinohio Research Services, Columbus, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - University of Pennsylvania-Perelman School of Medicine, Philadelphia, Pennsylvania
  - International Clinical Research Ic Research Murfreesboro, Murfreesboro, Tennessee
  - Arlington Center For Dermatology, Arlington, Texas
  - Austin Institute For Clinical Research Aicr Pflugerville, Pflugerville, Texas
  - University of Utah Health Care Midvalley Health Center Dermatology, Murray, Utah
- Canada (2):
  - Wiseman Dermatology Research Inc, Winnipeg, Manitoba
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 19 study centers in Canada and the United States.
Groups:
- Double-Blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 16 weeks.
- Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID: Participants applied matching vehicle cream BID for 16 weeks.
- Open-Label Extension (OLE) Period: Ruxolitinib Cream 1.5% BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week Open-label Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-blind, Vehicle-controlled Period continued to apply ruxolitinib cream 1.5% BID for an additional 16 weeks in the Open-label Extension Period.
- Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week Open-label Extension Period. Participants who applied vehicle cream BID during the Double-blind, Vehicle-controlled Period applied ruxolitinib cream 1.5% BID for 16 weeks in the Open-label Extension Period.
Period: 16-Week DBVC Period
Arm/Group | Double-Blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID | Open-Label Extension (OLE) Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 32 | 32 | 0 | 0
Completed | 30 | 29 | 0 | 0
Not Completed | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Period: 16-Week OLE Period
Arm/Group | Double-Blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID | Open-Label Extension (OLE) Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Started | 0 | 0 | 30 | 29
Completed | 0 | 0 | 29 | 23
Not Completed | 0 | 0 | 1 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (14.35) | 58.2 (10.86) | 57.3 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 21 | 19 | 40
  Black/African-American | 9 | 9 | 18
  Asian | 2 | 2 | 4
  Biracial | 0 | 1 | 1
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment-Treatment Success (IGA-TS) at Week 16
Description: The Investigator's Global Assessment (IGA) is a modified global assessment tool to assess the severity of lesions. Grading was based on 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), and 4 (severe). IGA-TS response was defined as an IGA score of 0 or 1 with a ≥2-grade improvement from Baseline at Week 16.
Time Frame: Baseline; Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups were defined according to the treatment assignment at the time of randomization regardless of the actual study drug the participant might have taken during their participation in the Double-blind; vehicle-controlled (DBVC) period. Missing post-Baseline values were imputed as nonresponders. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 32 | 32
percentage of participants | 50.0 [31.9 to 68.1] | 21.9 [9.3 to 40.0]
Statistical Analysis 1: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Superiority; p = 0.0129, Cochran-Mantel-Haenszel — stratified by Baseline Investigator's Global Assessment (IGA) score (3 or 4); Response Rate Difference = 29.4, 95% CI 2-sided [7.55 to 51.33], Standard Error of Mean 11.17 — stratified by Baseline IGA score (3 or 4)
Statistical Analysis 2: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Superiority; Odds Ratio (OR) = 4.04, 95% CI 2-sided [1.32 to 12.38] — stratified by Baseline IGA score (3 or 4)

2. Secondary Outcome: Percentage of Participants Achieving IGA-TS at Each Scheduled Post-Baseline Visit in the Double-Blind, Vehicle-Controlled Period
Description: The IGA is a global assessment tool to assess the severity of lesions. The IGA includes items such as depigmentation/hypopigmentation, lichenification (fine wrinkling/cigarette paper skin), excoriations, petechiae/ecchymosis, telangiectasias, erosions, fissures, or ulcers. Grading was based on 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), and 4 (severe). IGA-TS response was defined as an IGA score of 0 or 1 with a ≥2-grade improvement from Baseline at each scheduled post-Baseline visit. Participants with a score of 0 have a morphology of: no inflammatory signs (no erythema, no induration/papulation). Postinflammatory hyperpigmentation and/or hypopigmentation may be present. Participants with a score of 1 have a morphology of: barely perceptible erythema, barely perceptible induration/papulation/elevation, and/or minimal scale. Features include palpable, slightly erythematous papules.
Time Frame: Baseline; Weeks 2, 4, 8, 12, and 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 31
percentage of participants
  Week 2 | 9.7 [2.0 to 25.8] | 6.5 [0.8 to 21.4]
  Week 4: number analyzed (Participants) | 31 | 30
  Week 4 | 25.8 [11.9 to 44.6] | 13.3 [3.8 to 30.7]
  Week 8 | 51.6 [33.1 to 69.8] | 12.9 [3.6 to 29.8]
  Week 12: number analyzed (Participants) | 30 | 29
  Week 12 | 53.3 [34.3 to 71.7] | 24.1 [10.3 to 43.5]
  Week 16: number analyzed (Participants) | 30 | 29
  Week 16 | 53.3 [34.3 to 71.7] | 24.1 [10.3 to 43.5]
Statistical Analysis 1: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Equivalence — A Cochran-Mantel-Haenszel test stratified by Baseline IGA score (3 or 4) at a 2-sided α = 0.05 level was used for the comparison between ruxolitinib 1.5% cream BID and vehicle cream BID at Week 16; p = 0.0141, Cochran-Mantel-Haenszel; stratified by Baseline IGA score (3 or 4); Response Rate Difference = 30.6, 95% CI 2-sided [7.71 to 53.51], Standard Error of Mean 11.68
Statistical Analysis 2: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.16, 95% CI 2-sided [1.31 to 13.17] — stratified by Baseline IGA score (3 or 4)

3. Secondary Outcome: Percentage of Participants Achieving IGA-TS at Each Scheduled Post-Baseline Visit in the Open-label Extension Period
Description: as for outcome 2
Time Frame: Baseline; Weeks 18, 20, 24, 28, and 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Open-Label Extension Period: Ruxolitinib Cream 1.5% BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week Open-label Extension Period. Participants who applied ruxolitinib cream 1.5% BID during the Double-blind, Vehicle-controlled Period continued to apply ruxolitinib cream 1.5% BID for an additional 16 weeks in the Open-label Extension Period.
Arm/Group | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 30 | 28
percentage of participants
  Week 18: number analyzed (Participants) | 29 | 28
  Week 18 | 58.6 [38.9 to 76.5] | 25.0 [10.7 to 44.9]
  Week 20: number analyzed (Participants) | 29 | 27
  Week 20 | 62.1 [42.3 to 79.3] | 33.3 [16.5 to 54.0]
  Week 24: number analyzed (Participants) | 29 | 25
  Week 24 | 58.6 [38.9 to 76.5] | 44.0 [24.4 to 65.1]
  Week 28: number analyzed (Participants) | 29 | 24
  Week 28 | 58.6 [38.9 to 76.5] | 45.8 [25.6 to 67.2]
  Week 32: number analyzed (Participants) | 30 | 23
  Week 32 | 60.0 [40.6 to 77.3] | 60.9 [38.5 to 80.3]

4. Secondary Outcome: Percentage of Participants With ITCH4 at Each Scheduled Post-Baseline Visit in the Double-Blind, Vehicle-Controlled Period
Description: ITCH4 response was defined as a ≥4-point improvement in the Itch Numeric Rating Scale (NRS) score from Baseline at each scheduled post-Baseline visit, up to and including Week 32. The Itch NRS is a daily participant-reported measure (24-hour recall) of the worst level of itch intensity. Participants were instructed to complete and record their Itch NRS in a diary each evening beginning on the day of screening through Week 32 or treatment discontinuation. Participants rated itch severity of their lichen planus by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best described the worst level of itch they experienced in the past 24 hours.
Time Frame: Baseline; Weeks 2, 4, 8, 12, and 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 29 | 30
percentage of participants
  Week 2: number analyzed (Participants) | 28 | 30
  Week 2 | 21.4 [8.3 to 41.0] | 3.3 [0.1 to 17.2]
  Week 4: number analyzed (Participants) | 29 | 28
  Week 4 | 44.8 [26.4 to 64.3] | 7.1 [0.9 to 23.5]
  Week 8: number analyzed (Participants) | 26 | 27
  Week 8 | 53.8 [33.4 to 73.4] | 7.4 [0.9 to 24.3]
  Week 12: number analyzed (Participants) | 25 | 25
  Week 12 | 52.0 [31.3 to 72.2] | 12.0 [2.5 to 31.2]
  Week 16: number analyzed (Participants) | 26 | 26
  Week 16 | 57.7 [36.9 to 76.6] | 19.2 [6.6 to 39.4]
Statistical Analysis 1: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0027, Cochran-Mantel-Haenszel; stratified by Baseline IGA score (3 or 4); Response Rate Difference = 40.3, 95% CI 2-sided [16.61 to 64.00], Standard Error of Mean 12.09
Statistical Analysis 2: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 6.67, 95% CI 2-sided [1.85 to 24.02] — stratified by Baseline IGA score (3 or 4)

5. Secondary Outcome: Percentage of Participants With ITCH4 at Each Scheduled Post-Baseline Visit in the Open-label Extension Period
Description: as for outcome 4
Time Frame: Baseline; Weeks 18, 20, 24, 28, and 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 24 | 25
percentage of participants
  Week 18: number analyzed (Participants) | 22 | 25
  Week 18 | 72.7 [49.8 to 89.3] | 48.0 [27.8 to 68.7]
  Week 20: number analyzed (Participants) | 23 | 22
  Week 20 | 73.9 [51.6 to 89.8] | 63.6 [40.7 to 82.8]
  Week 24: number analyzed (Participants) | 24 | 21
  Week 24 | 79.2 [57.8 to 92.9] | 76.2 [52.8 to 91.8]
  Week 28: number analyzed (Participants) | 22 | 17
  Week 28 | 86.4 [65.1 to 97.1] | 76.5 [50.1 to 93.2]
  Week 32: number analyzed (Participants) | 19 | 15
  Week 32 | 84.2 [60.4 to 96.6] | 73.3 [44.9 to 92.2]

6. Secondary Outcome: Time to Achieve ITCH4 in the Double-blind, Vehicle-controlled Period
Description: as for outcome 4
Time Frame: up to Week 16
Population: ITT Population. Only those participants achieving a ≥4-point improvement in daily Itch NRS score from Baseline were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 32 | 31
days | 17.0 [7.0 to 27.0] | 97.0 [31.0 to NA] — The upper limit of the confidence interval was not estimable because there were too few events of ITCH4 response.
Statistical Analysis 1: Comparison: Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID vs Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID; Test type: Equivalence — A log-rank test stratified by randomization stratification factor, Baseline IGA score (3 or 4), was used for between-treatment group comparisons. The hazard ratio and its 95% confidence interval was estimated based on the stratified Cox regression model. using Efron's method accounting for ties; p = 0.0008, Log Rank; stratified by Baseline IGA score (3 or 4) between ruxolitinib 1.5% cream and vehicle cream; Hazard Ratio (HR) = 2.850, 95% CI 2-sided [1.510 to 5.381] — Cox regression model stratified by Baseline IGA score (3 or 4) was conducted to compare the difference in hazard rate between ruxolitinib 1.5% cream and vehicle cream

7. Secondary Outcome: Change From Baseline in the Skin Pain NRS Score at Each Scheduled Post-Baseline Visit in the Double-Blind, Vehicle-Controlled Period
Description: Participants were instructed to complete and record the Skin Pain NRS in a diary each evening beginning on the day of screening through Week 32 or treatment discontinuation. Participants rated their pain, which included all types of pain (e.g., burning, tearing, pulling, stabbing, etc.) severity of lichen planus by selecting a number from 0 (no pain) to 10 (worst imaginable pain) that best described the worst level of pain they experienced in the past 24 hours. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 2, 4, 8, 12, and 16
Population: ITT Population. No imputation was performed for missing values. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 31
scores on a scale
  Baseline | 4.86 (2.303) | 4.51 (2.618)
  Week 2: number analyzed (Participants) | 28 | 30
  Week 2 | -1.69 (2.047) | -0.55 (0.975)
  Week 4: number analyzed (Participants) | 29 | 28
  Week 4 | -2.64 (2.307) | -0.69 (1.261)
  Week 8: number analyzed (Participants) | 26 | 27
  Week 8 | -2.96 (2.622) | -0.95 (1.385)
  Week 12: number analyzed (Participants) | 25 | 25
  Week 12 | -3.01 (2.823) | -0.84 (1.613)
  Week 16: number analyzed (Participants) | 26 | 26
  Week 16 | -3.02 (2.656) | -1.25 (2.263)

8. Secondary Outcome: Change From Baseline in the Skin Pain NRS Score at Each Scheduled Post-Baseline Visit in the Open-label Extension Period
Description: as for outcome 7
Time Frame: Baseline; Weeks 18, 20, 24, 28, and 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 31 | 31
scores on a scale
  Baseline | 4.86 (2.303) | 4.51 (2.618)
  Week 18: number analyzed (Participants) | 22 | 25
  Week 18 | -3.65 (2.086) | -2.46 (2.253)
  Week 20: number analyzed (Participants) | 23 | 22
  Week 20 | -3.81 (2.079) | -2.96 (2.584)
  Week 24: number analyzed (Participants) | 24 | 21
  Week 24 | -3.82 (2.385) | -3.13 (2.868)
  Week 28: number analyzed (Participants) | 22 | 17
  Week 28 | -3.99 (2.272) | -3.54 (3.145)
  Week 32: number analyzed (Participants) | 19 | 16
  Week 32 | -4.25 (2.276) | -3.51 (3.470)

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) During the Double-blind, Vehicle-controlled Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from Baseline to Week 16 plus 30 days
Population: Safety Population: all participants who applied ruxolitinib 1.5% cream BID or vehicle cream BID at least once. Treatment groups for this population were determined according to the actual treatment the participant applied on Day 1 regardless of assigned study drug treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 32
Participants | 15 | 9

10. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE During the Double-blind, Vehicle-controlled Period
Description: A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of AEs was assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v5.0) Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to 1 of the following categories: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: from Baseline to Week 16 plus 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind, Vehicle-Controlled Period: Ruxolitinib Cream 1.5% BID | Double-Blind, Vehicle-Controlled Period: Vehicle Cream BID
Number analyzed (Participants) | 31 | 32
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Any TEAE During the Open-label Extension Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from Week 17 to Week 32 plus 30 days
Population: Open-label Extension Evaluable Population: all participants who applied ruxolitinib 1.5% cream at least once during the Open-label Extension Period
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 30 | 29
Participants | 8 | 11

12. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE During the Open-label Extension Period
Description: A TEAE was defined as an AE either reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of AEs was assessed using the CTCAE v5.0 Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to 1 of the following categories: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: from Week 17 to Week 32 plus 30 days
Population: Open-label Extension Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Extension Period: Ruxolitinib Cream 1.5% BID | Open-Label Extension Period: Vehicle Cream to Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 30 | 29
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: from Baseline to Week 32 plus 30 days
Description: For safety analysis, participants who switched from treatment with vehicle to treatment with ruxolitinib cream 1.5% BID in the Open-Label Extension Period have been counted both in the vehicle arm and the ruxolitinib arm.
Groups:
- Vehicle Cream BID: Participants applied matching vehicle cream BID for 16 weeks in the Double-Blind, Vehicle-Controlled Period.
- Ruxolitinib Cream 1.5% BID: Participants who applied ruxolitinib cream 1.5% BID for 16 weeks during the Double-Blind, Vehicle-Controlled Period plus participants who completed the Week 16 assessments with no safety concerns, continued into the Open-label Extension Period, and applied ruxolitinib cream 1.5% BID for an additional 16 weeks
Arm/Group | Vehicle Cream BID | Ruxolitinib Cream 1.5% BID
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/60
Other Adverse Events (participants affected / at risk) | 6/32 | 14/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=32) | Ruxolitinib Cream 1.5% BID (N=60)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT05593432/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05593432/SAP_001.pdf